CLINICAL TRIAL: NCT04572932
Title: Evaluation of the Use of Probiotics In Patients With Irritable Bowel Syndrome
Brief Title: Probiotics and Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate Professor of Tropical Medicine, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Irritable Bowel Syndrome
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: intestinal microbiota,; probiotics,; quality of life,
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1:Probiotic arm (Active Comparator): first group was prescribed probiotics (10 billion colony of lactobacillus delbruekii and lactobacillus fermentum) and itopride hcl 50mg three times daily for 4 weeks
  Interventions: Drug: lactobacillus delbruekii
- Group 2:Placcebo arm (Active Comparator): the second group received only itopridehcl 50mg by the same dose for four weeks.
  Interventions: Drug: lactobacillus delbruekii

INTERVENTIONS:
Drug: lactobacillus delbruekii — Comarsion between probiotics and one of the most widely used symptomatc treatment for IBS itopride hcl
  Other Names: and lactobacillus fermentum); and itopride hcl

SUMMARY:
This clinical trial was conducted on 90 IBS patients, who fulfill ROME IV criteria and the IBS diagnostic questionnaire (Arabic version licensed by Rome Foundation) in Egyptair hospital outpatient clinic, Cairo, Egypt between May and December 2019. Data of the patient, with suspected IBS during the study period, were reviewed and the patients who fulfilled the inclusion criteria were enrolled into this study. A written consent was obtained from all included patients. The patients who agreed to participate were then randomly assigned into two equal groups and were followed up after 4 weeks from the first visit.

DETAILED DESCRIPTION:
The study includes 90 patients assigned into2 equal groups the first was prescribed probiotics (10 billion colony of lactobacillus delbruekii and lactobacillus fermentum) and itopride hcl 50mg three times daily, while the second group receivedonly itopridehcl 50mg by the same dose for four weeks.All patients fulfill ROME IV criteria and the IBS diagnostic questionnaire (Arabic version licensed by Rome Foundation). Data of the patient, with suspected IBS during the study period, were reviewed and the patients who fulfilled the inclusion criteria were enrolled into this study. A written consent was obtained from all included patients. The patients who agreed to participate were then randomly assigned into two equal groups and were followed up after 4 weeks from the first visit.

Any patient with red flags (e.g. weight or appetite loss, iron deficiency anemia, fever or rectal bleeding), Known inflammatory bowel disease or celiac disease patients, patients above 50 years of age and immuno-compromised patients were excluded from the study.

The included patients aged from 18 to 50 years fulfilling Rome IV criteria for diagnosis of IBS:Recurrent abdominal pain (on average, at least 1 day/week in the last 3 months) associated with two or more of the following: (Related to defecation, Associated with a change in frequency of stool, Associated with a change in form of stool).Patients should fulfill Rome Foundation IBS-Diagnostic Questionnaire.

All patients were subjected to initial evaluation byfull history taking, questionnaires for (IBS diagnostic questionnaire, IBS-SSSand QOL -IBS survey), clinical examination, investigations (including CBC, ESR, CRP, random sugar, HbA1c, thyroid profile and stool analysis) and radiological assessment bypelvi-abdominal ultrasound to exclude any organic cause..Group one(45 patients) was prescribed probiotic (lactobacillus delbruekii and l. fermentum) 10billion colony forming units and itopride 50mg three times daily for four weeks while group two was prescribed only itopride 50mg three times daily for four weeks.Then reassessment of the questionnaires was done after 4 weeks of treatment for comparison

ELIGIBILITY:
Inclusion Criteria:

1-Patients should fulfill Rome Foundation IBS-Diagnostic Questionnaire i.e [Recurrent abdominal pain (on average, at least 1 day/week in the last 3 months) associated with two or more of the following: (Related to defecation, Associated with a change in frequency of stool, Associated with a change in form of stool)].

Exclusion Criteria:

1. Any patient with red flags (e.g. weight or appetite loss, iron deficiency anemia, fever or rectal bleeding),
2. Known inflammatory bowel disease or celiac disease patients,
3. patients above 50 years of age
4. immuno-compromised patients
5. Refusal to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Change of IBS Symptoms | 4 weeks
  via Irritable bowel syndrom severity scale (IBS-SSS Arabic version)

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
To publish the results of this research . further studies on larger number of patients and for longer durtion as future plan